CLINICAL TRIAL: NCT07002658
Title: Endoscopic Saphenous Vein Harvesting Versus Conventional Open Harvesting in Patients Undergoing Coronary Artery Bypass Grafting, Either Alone or in Combination With Another Cardiac Surgical Procedure, in Terms of the Clinical Impact of Surgical Wound Morbidity
Brief Title: Clinical Impact of Surgical Wound Morbidity According to the Type of Saphenous Vein Harvesting Technique (Endoscopic vs. Open) in Patients Undergoing Myocardial Revascularization Surgery
Acronym: EndOSiC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, María Belén Solís Chávez, Cardiac Surgery Resident, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25/148-E
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: CABG-patients; Saphenectomy; Endoscopic Surgery; Wound Complications; Antibiotic Use; Cardiac Surgery; Off Pump Coronary Artery Bypass Graft; Coronary Artery Bypass Graft With or Without ECC
Keywords: endoscopic vein harvesting; CABG surgery; open vein harvesting; wound morbidity

STUDY DESIGN:
Intervention Model Description: One group will receive the open technique for saphenous vein harvesting and the other group will receive the endoscopic technique.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic saphenectomy (Experimental): Endoscopic vein harvesting in CABG surgery requiring a vein graft with or without extracorporeal circulation
  Interventions: Procedure: Harvesting of the saphenous vein graft
- Conventional and open technique for saphenous vein harvesting (Active Comparator): Using the conventional open technique for harvesting the saphenous vein in any type of surgery with or without extracorporeal circulation
  Interventions: Procedure: Harvesting of the saphenous vein graft

INTERVENTIONS:
Procedure: Harvesting of the saphenous vein graft — Most existing studies on endoscopic saphenectomy have been conducted in CABG with cardiopulmonary bypass (CBP), whereas most CABG surgeries at the study center are performed without CBP.
  The following outcomes will be identified:
  * Days of admission or need for hospitalization
  * Use of antibiotic therapy for saphenectomy wound infections
  * Need for wound dressings due to necrosis and/or wound infection
  * Need for analgesic treatment for wound pain

SUMMARY:
The goal of this clinical trial is to compare two different techniques: endoscopic saphenous vein harvesting versus conventional open harvesting in patients undergoing coronary artery bypass grafting, either alone or in combination with another cardiac surgical procedure (valve surgery or arrhythmia surgery). The main questions the trial aims to answer are:

Does the endoscopic technique reduce surgical wound morbidity in terms of shorter hospital stays? Does endoscopic saphenous harvesting reduce the use of antibiotics for saphenectomy wound infections? Does the endoscopic technique reduce need for wound dressings due to necrosis and/or wound infection, and reduce need for analgesic treatment for wound pain? This prospective, randomized study will be conducted in the Cardiovascular Surgery Service at Hospital Clínico San Carlos.

Participants will be randomly assigned to a different saphenectomy technique. All patients will be assessed for saphenectomy wound complications upon discharge, and by phone call at 7 days, 1 month, and 3 months following the intervention.

DETAILED DESCRIPTION:
* Pain in the leg incisions will be assessed using a standarized pain scale.
* Antibiotic and analgesic requirements for infection or pain in the saphenous vein surgical wound will be documeted.
* The need for outpatient treatment or hospitalization due to surgical wounds will be evaluated.
* A surgical wound cosmetic satisfaction survey will be administered to participants.

  * Images of the saphenectomy surgical wound will be collected at 1 month postoperatively.
  * Major cardiovascular events will be monitored during follow-up visits or hospital admissions and recorded in the RECC database (local service database)

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary artery bypass grafting (CABG), alone or in combination with other surgery (valve or arrhythmia surgery), with or without cardiopulmonary bypass (CPB), in which preoperative evaluation includes the plan to use a short saphenous vein segment (alone or in addition to arterial conduits).
* Availability of a surgeon or cardiac surgery resident trained in endoscopic harvesting in the operating room.
* Patients undergoing myocardial revascularization surgeries with or without extracorporeal circulation.
* Patients undergoing concomitant cardiac valve replacement surgery, atrial fibrillation surgery, and others, in addition to CABG

Exclusion Criteria:

* Emergent surgery or procedures performed during cardiorespiratory arrest
* Myocardial revascularization with arterial grafts only
* Presence of varicose veins
* History of infrainguinal vascular surgery
* Presence of ulcers and/or active infection in the lower limbs
* Previous stroke with neurological sequelae in the legs
* History of deep vein thrombosis in the legs
* Pregnancy
* Age under 18 years
* Lack of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Wound morbidity | From enrollment to the three-month follow-up visit
  Days of hospital stay, use of antibiotics for saphenectomy wound infections, need for wound dressings due to necrosis and/or wound infection, and need for analgesic treatment for wound pain.
  1. Length of Hospital Stay. Unit of Measure: Days
  2. Use of Antibiotics for Saphenectomy Wound Infections Measure: Number of participants requiring oral or parenteral antibiotics due to wound infection. Unit of Measure: Participants
  3. Need for Wound Dressings Due to Necrosis and/or Infection Measure: Number of participants requiring wound dressings due to necrosis and/or wound infection. Unit of Measure: Participants
  4. Use of Analgesics for Wound Pain Measure: Number of participants requiring analgesic treatment for saphenectomy wound pain

SECONDARY OUTCOMES:
Freedom from combined cardiac events | 1 year
  Freedom from death, myocardial infarction, and recurrent angina

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Clínico San Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
the IPD data will be share at the end of the study

REFERENCES:
- [Background] Zenati MA, Bhatt DL, Bakaeen FG, Stock EM, Biswas K, Gaziano JM, Kelly RF, Tseng EE, Bitondo J, Quin JA, Almassi GH, Haime M, Hattler B, DeMatt E, Scrymgeour A, Huang GD; REGROUP Trial Investigators. Randomized Trial of Endoscopic or Open Vein-Graft Harvesting for Coronary-Artery Bypass. N Engl J Med. 2019 Jan 10;380(2):132-141. doi: 10.1056/NEJMoa1812390. Epub 2018 Nov 11. PMID 30417737
- [Background] Sousa-Uva M, Neumann FJ, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur J Cardiothorac Surg. 2019 Jan 1;55(1):4-90. doi: 10.1093/ejcts/ezy289. No abstract available. PMID 30165632
- [Background] Sampath HK, Lee TJH, Cher CE, Liang S, Cheong OO, Kofidis T, Vitaly S, Sazzad F. A Comprehensive Clinical Outcome Analysis of Endoscopic Vessel Harvesting for Coronary Artery Bypass Surgery. J Clin Med. 2024 Jun 11;13(12):3405. doi: 10.3390/jcm13123405. PMID 38929933
- [Background] Li G, Zhang Y, Wu Z, Liu Z, Zheng J. Mid-term and long-term outcomes of endoscopic versus open vein harvesting for coronary artery bypass: A systematic review and meta-analysis. Int J Surg. 2019 Dec;72:167-173. doi: 10.1016/j.ijsu.2019.11.003. Epub 2019 Nov 9. PMID 31707009
- [Background] Kopjar T, Dashwood MR. Towards Endoscopic No-Touch Saphenous Vein Graft Harvesting in Coronary Bypass Surgery. Braz J Cardiovasc Surg. 2022 Sep 2;37(Spec 1):57-65. doi: 10.21470/1678-9741-2022-0144. PMID 36054003
- [Background] Kodia K, Patel S, Weber MP, Luc JGY, Choi JH, Maynes EJ, Rizvi SA, Horan DP, Massey HT, Entwistle JW, Morris RJ, Tchantchaleishvili V. Graft patency after open versus endoscopic saphenous vein harvest in coronary artery bypass grafting surgery: a systematic review and meta-analysis. Ann Cardiothorac Surg. 2018 Sep;7(5):586-597. doi: 10.21037/acs.2018.07.05. PMID 30505742
- [Background] Fudulu D, Angelini GD. Saphenous vein graft longevity: open or endoscopic, with VEST or without? Eur J Cardiothorac Surg. 2022 Jun 15;62(1):ezac144. doi: 10.1093/ejcts/ezac144. No abstract available. PMID 35323908
- [Background] Allen KB, Heimansohn DA, Robison RJ, Schier JJ, Griffith GL, Fitzgerald EB. Influence of endoscopic versus traditional saphenectomy on event-free survival: five-year follow-up of a prospective randomized trial. Heart Surg Forum. 2003;6(6):E143-5. PMID 14722001